CLINICAL TRIAL: NCT01995006
Title: Effect of Metamizole on Renal Function in Salt-depleted Healthy Subjects Single-center, Randomized, Open, Controlled Parallel-group Study to Investigate the Effects of Oral Metamizole or Naproxen on Renal Function in Healthy Male Salt-depleted Subjects
Brief Title: Effect of Metamizole (Dipyrone) on Renal Function in Salt-depleted Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EKBB 264/13
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: Effect; metamizole; salt-depleted; subjects
MeSH Terms: interventions — Dipyrone; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metamizole (Experimental): Metamizole 1000mg TID Day 1 till Day 7
  Interventions: Drug: metamizole
- Naproxen (Active Comparator): Naproxen 500 mg BID Day 1 till Day 7
  Interventions: Drug: Naproxen

INTERVENTIONS:
Drug: metamizole — metamizol tablets (500mg): 1000mg TID during 7 days
  Other Names: dipyrone
  Arms: Metamizole
Drug: Naproxen — Naproxen tablets (500mg): 500 mg BID during 7 days
  Other Names: Naproxen sodium
  Arms: Naproxen

SUMMARY:
The planned study is a single-center, randomized, open-label parallel group study in 16 healthy male subjects. Study subjects will be randomly allocated either to the metamizole group (1) or to the naproxen group (2). All participants will start with a low sodium diet (approximately 50 mmol Na+ per day) 7 days before the first drug intake and maintain the diet until the end of the study (14 days in total). Salt-depletion is an accepted model to enhance production of vasodilatory prostaglandins and to increase renal sensitivity to prostaglandin inhibition. On the first day of treatment (Day 1), a single dose of metamizole or naproxen will be administered to investigate the effects after a single dose and to collect single dose pharmacokinetic profiles. Starting on Day 2, all participants will receive therapeutic doses, i.e. 1000 mg metamizole 'ter in die' (TID, three times a day) or 500 mg naproxen 'bis in die' (BID, twice a day) for one week and on Day 7 pharmacokinetics and pharmacodynamics effects will be assessed under near steady-state conditions.

The primary objective is the characterization of the renal effects of metamizole by determination of the glomerular filtration rate (GFR) using the inulin clearance. Secondary objectives are the characterization of the urinary excretion of prostaglandin E2 (PGE2) and the prostaglandin I2 (PGI2) metabolite 6-keto-prostaglandin F1 (PGF1)alpha as well as the urinary excretion of sodium and potassium.

Overall, clinical experience suggests better renal tolerability of metamizole possibly due to less potent COX-inhibition compared to classical nonsteroidal antiinflammatory drugs (NSAIDs). If this could be confirmed, metamizole would be a valuable alternative for treatment of painful conditions in patients with impaired renal function. Therefore, the aim of this study is to examine the effects of metamizole on renal function in comparison with the non-specific COX-inhibitor naproxen.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged between 18 and 45 years (inclusive) at screening
* BMI between 18 and 28 kg/m2 (inclusive) and body weight at least 50 kg at screening.
* systolic blood pressure (SBP): 100-140 mmHg, diastolic blood pressure (DBP): 60-90 mmHg and heart rate (HR): 45-90 bpm (inclusive), measured on the leading arm*, in the supine position at screening.
* No clinically significant findings on the physical examination at screening.
* 12-lead ECG without clinically relevant abnormalities at screening.
* Signed informed consent prior to any study-mandated procedure.
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening.
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study.

  * leading arm right = writing with right hand

Exclusion Criteria:

* Smoking > 5 cigarettes per day.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Loss of ≥ 250 ml of blood within 3 months prior to screening.
* Treatment with an investigational drug within 30 days prior to screening.
* Previous treatment with any prescribed or over-the-counter (OTC) medication (including herbal medicines such as St John's Wort) within 2 weeks prior to the intended start of the study.
* Legal incapacity or limited legal capacity at screening.
* Positive results from urine drug screen at screening.
* History or clinical evidence of any disease (e.g. GIT-disease: Morbus Crohn, Colitis Ulcerosa, anamnestic gastrointestinal bleeding) and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk for toxicity.
* Known hypersensitivity to Aspirin or other NSAIDs or any excipients of the drug formulations.
* Known food allergy, which make the adherence to the diet impossible
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (GFR) | up to 7 days

SECONDARY OUTCOMES:
Measurement of the urinary excretion of the prostaglandin E2 (PGE2) and of the prostacyclin (PGI2) metabolite 6-keto-PGF1alpha | Day 1 and Day 7
Measurement of urine levels of sodium, potassium and creatinine and the urinary output | Day 1 and Day 7
Plasma pharmacokinetic (PK) parameters of each drug will be derived either directly from observed data or by analysis of the concentration-time profiles | Day 1 and Day 7
  * The maximum plasma concentration (Cmax) and time to reach Cmax (tmax)
  * The terminal elimination rate constant with the respective half-life (t½)
  * The area under the plasma concentration-time curve from zero to different time points (AUC0-24, AUC0-∞)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Haschke, PD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Phase I Research Unit, University Hospital, Basel, Switzerland